CLINICAL TRIAL: NCT05102825
Title: Imaging Measures of Respiratory Health Registry
Acronym: iMRH
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Rayment, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H19-01163
Record Dates: First submitted 2021-09-27; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Disease; Healthy
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Respiratory Disease: Any physician-diagnosed lung disease
  Interventions: Diagnostic Test: 1H and Xe-129 MRI
- Healthy: Healthy control with no physician-diagnosed lung disease
  Interventions: Diagnostic Test: 1H and Xe-129 MRI

INTERVENTIONS:
Diagnostic Test: 1H and Xe-129 MRI — Traditional 1H-MRI (room air inhalation) and Xe-129 MRI (requires inhalation of Xenon 129 gas).

SUMMARY:
This is a prospective, observational cohort registry that aims to collect data on pulmonary structure and function in healthy people and those with respiratory disease, using structural and functional pulmonary 1H-MRI and hyperpolarized 129Xe-MRI.

Outcome measures generated from MRI may include but are not limited to measures of regional ventilation, pulmonary microarchitecture, and regional gas exchange. Additionally, one of the goals of the registry is to facilitate the development of novel image analysis techniques that have not yet been invented.

These data will be stored along with demographic data, clinical data, and pulmonary function testing (PFT) data.

This is an open registry. Eligible local and international investigators/institutions can apply for access.

ELIGIBILITY:
Respiratory Disease

Inclusion Criteria:

1. Physician-diagnosed lung disease - based on a diagnosis made by a treating staff physician and confirmed by the principal investigator.
2. Age 0-99 years.
3. Informed consent by participant, parent, or legal guardian
4. In the opinion of the Investigator, the participant will likely be able to perform maneuvers to obtain technically acceptable pulmonary XeMRI images.

Exclusion Criteria:

1. Physical findings at screening that, in the opinion of the Investigator, would compromise the safety of the participant or the quality of the research data.
2. Requirement of supplementary oxygen to maintain an oxygen saturation above 95%.
3. Failed MRI screening form.
4. History of claustrophobia.
5. Known current pregnancy or lactation.

Healthy

Inclusion Criteria:

1. Age 0-99 years
2. Informed consent by participant, parent, or legal guardian
3. In the opinion of the Investigator, the participant will likely be able to perform maneuvers to obtain technically acceptable pulmonary MRI images.

Exclusion Criteria

1. Physician-diagnosed lung disease.
2. Failed MRI screening form.
3. History of claustrophobia.
4. Physical findings at screening that, in the opinion of the Investigator, would compromise the safety of the participant or the quality of the research data.
5. Known current pregnancy or lactation.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible individuals with respiratory disease will be identified from various Respiratory Medicine or subspecialty clinics at British Columbia Children's Hospital (BCCH) or from analogous clinics at St Paul's Hospital (SPH). Participants may be contacted using a First Contact Letter, or permission to approach will be obtained by a member of their circle of care.
  Healthy participants will be recruited from family members of patients in the Division of Respiratory Medicine at BCCH and SPH as well as from the community or other clinics using flyers or a First Contact Letter.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2045-06-01 (Estimated); Study Completion 2045-06-01 (Estimated)

PRIMARY OUTCOMES:
Structural proton (1H) MRI data | no predefined schedule in this open registry study; maximum 25 visits, over up to 25 years
  Includes all proton MRI images collected to assess pulmonary structure. Data may be analysed qualitatively and quantitatively.
Functional proton (1H) MRI data | no predefined schedule in this open registry study; maximum 25 visits, over up to 25 years
  Includes all proton MRI images collected to assess pulmonary function. Data may be analysed qualitatively and quantitatively.
Functional hyperpolarized 129-xenon (129Xe) MRI data | no predefined schedule in this open registry study; maximum 25 visits, over up to 25 years
  Includes all proton images collected to assess pulmonary function. Data may be analysed qualitatively and quantitatively.

SECONDARY OUTCOMES:
Resting oxygen saturation | no predefined schedule in this open registry study; maximum 25 visits, over up to 25 years
CFQ-R Respiratory domain | no predefined schedule in this open registry study; maximum 25 visits, over up to 25 years
  Only for participants with cystic fibrosis
St. George Respiratory Questionnaire | no predefined schedule in this open registry study; maximum 25 visits, over up to 25 years
  Only for participants with Respiratory disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rayment, MDCM, MSc, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
iMRH-Registry Data may be shared with investigators from BCCHR/UBC or elsewhere. iMRH-Registry Co-Investigaotrs using iMRH Registry Data to address the Scientific Objectives of the iMRH Registry do not need to formally apply for access. All other User-Investigators (domestic and international) must apply to the iMRH-Registry Data Access Committee for access to the iMRH-Registry Data.
Access Criteria: Criteria for access to the iMRH-Registry Data:
  1. The Proposed Study must demonstrate approval by a Qualified REB
  2. The objectives of the Proposed Study must align with the scientific objectives of the iMRH-Registry (see §5)
  3. Use of the iMRH Registry Data in the Proposed Study must respect the informed consent given by the participants of the iMRH Registry;
  4. The Proposed Study must have scientific merit, as assessed by the iMRH Registry Data Access Committee
  5. The User-Investigator must demonstrate sufficient funding to perform the Proposed Study.